CLINICAL TRIAL: NCT01218841
Title: Clinical and Immunological Benefits of the Infusion of Pure Fish Oil Lipid Emulsion in Surgical Patients With Gastrointestinal Cancer.
Brief Title: Pure Fish Oil Parenteral Lipid Emulsion in Patients With Gastrointestinal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Dan Linetzky Waitzberg - Professor, University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAPPesq 310/04
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2010-10

CONDITIONS: Surgery
Keywords: Fish oil; Omega-3 fatty acids; Parenteral lipid emulsions; Immune response; Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish oil lipid emulsion (Experimental): Parenteral lipid emulsion composed by fish oil which is rich in the omega-3 polyunsaturated fatty acids eicosapentanoic and docosahexanoic.
  Interventions: Dietary Supplement: Fish oil lipid emulsion
- MCT/LCT lipid emulsion (Active Comparator): Parenteral lipid emulsion containing 50% of medium-chain triglycerides and 50% of soybean oil
  Interventions: Dietary Supplement: MCT/LCT

INTERVENTIONS:
Dietary Supplement: Fish oil lipid emulsion — 0.2g of fat/kg of body weight/day for 3 days during 6 continuous hours in peripheral vein.
  Other Names: Omegavenos
  Arms: Fish oil lipid emulsion
Dietary Supplement: MCT/LCT — 0.2g of fat/kg of body weight/day for 3 days during 6 continuous hours in peripheral vein.
  Other Names: Lipovenos MCT
  Arms: MCT/LCT lipid emulsion

SUMMARY:
Surgical trauma can lead to an intense inflammation and impairment of the capacity to fight against infections. Fish oil is composed by substances called omega-3 fatty acids which have anti-inflammatory effects. When infused through the vein as part of a nutritional treatment of some surgical patients, fish oil have been shown to preserve some defense capabilities against infections and to decrease postoperative release of inflammatory substances, contributing to the shortening of length of hospital and intensive care unity (ICU) stay and complications, mainly infectious complications. These reported benefits have been encouraging the vein infusion of fish oil as a kind of medicine to contribute for the treatment of surgical patients. In current study the investigators evaluated the effect of preoperative infusion of pure fish oil in patients with gastrointestinal cancer (stomach and colon) on their clinical outcomes. The hypothesis considered that preoperative infusion of fish oil, not as part of nutritional therapy but as a medicine agent, can attenuates inflammation and improves the capacity of surgical patients to fight against infections, improving their treatment.

ELIGIBILITY:
Inclusion Criteria:

Elective surgical patients with confirmed (biopsy) gastrointestinal (colon or stomach) cancer; 30-75 years old; venous assess to blood collections (40 mL) to receive parenteral infusions of lipid emulsion; Karnofsky performance statuses of ≥60

Exclusion Criteria:

Intolerance or allergy to any ingredient in lipid emulsion; diagnosis of infectious, inflammatory, immunologic or metabolic diseases; dementia;medicine intake that could significantly modulate metabolism; implanted electromagnetic instruments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2005-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan L. Waitzberg, PhD, Principal Investigator — University of Sao Paulo, Faculty of Medicine

REFERENCES:
- [Derived] de Miranda Torrinhas RS, Santana R, Garcia T, Cury-Boaventura MF, Sales MM, Curi R, Waitzberg DL. Parenteral fish oil as a pharmacological agent to modulate post-operative immune response: a randomized, double-blind, and controlled clinical trial in patients with gastrointestinal cancer. Clin Nutr. 2013 Aug;32(4):503-10. doi: 10.1016/j.clnu.2012.12.008. Epub 2012 Dec 22. PMID 23398953
- [Derived] Cury-Boaventura MF, Torrinhas RS, de Godoy AB, Curi R, Waitzberg DL. Human leukocyte death after a preoperative infusion of medium/long-chain triglyceride and fish oil parenteral emulsions: a randomized study in gastrointestinal cancer patients. JPEN J Parenter Enteral Nutr. 2012 Nov;36(6):677-84. doi: 10.1177/0148607111432759. Epub 2012 Jan 26. PMID 22282868